CLINICAL TRIAL: NCT04376359
Title: The Effectiveness of Hyperbaric Oxygen Therapy on Pneumonia Complicating
Brief Title: The Effectiveness of Hyperbaric Oxygen Therapy on Pneumonia Complicating Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ya Zhang (Other)
Responsible Party: Sponsor-Investigator, Ya Zhang, Principal Investigator, Anhui Medical University
Organization: Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018jyxm0772
Record Dates: First submitted 2020-05-03; First posted 2020-05-06 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Hyperbaric Oxygen Therapy; Stroke; Pneumonia
Keywords: Oral opportunistic pathogens; Pneumonia complicating stroke; Metagenome
MeSH Terms: conditions — Stroke; Pneumonia | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hyperbaric oxygen therapy (Experimental): Patients with stroke will receive the hyperbaric oxygen therapy (HBOT) for 40 times, which were completed on 40 business days over a 2-month period and each session lasted 90 minutes at 100% oxygen concentration and 2 atmospheres.
  Interventions: Procedure: hyperbaric oxygen therapy
- Control (No Intervention): Stroke patients were not treated with HBOT except for the same routine treatment as the experimental group.

INTERVENTIONS:
Procedure: hyperbaric oxygen therapy — Hyperbaric oxygen therapy is the patient put in airtight oxygen tank, by increasing the air pressure in the environment (1.5 to 3.0) under atmospheric pressure, to give 100% oxygen, the patient treatment time is approximately 60 minutes to 120 minutes in this way, can achieve the purpose of greatly increase the oxygen partial pressure in the organization, so as to achieve reverse brain edema, reduce lipid peroxidation, inhibiting leukocyte hyperactivity, rebuild the blood brain barrier.
  Arms: hyperbaric oxygen therapy

SUMMARY:
To investigate the evidence for the integration of hyperbaric oxygen therapy (HBOT) as part of interdisciplinary stroke rehabilitation.

DETAILED DESCRIPTION:
Pneumonia complicating stroke is very difficult to manage and has a very poor prognosis, leading to a significantly higher risk of death. Oral opportunistic pathogens have been reported to be associated with the incidence of pneumonia among non-stroke immunocompromised subjects. Preliminary studies found that patients with stroke had higher carriage rates of oral opportunistic pathogens than healthy subjects. Therefore, investigators hypothesize that pneumonia complicating stroke is associated with oral opportunistic pathogens, and hyperbaric oxygen therapy may reduce the incidence of pneumonia complicating stroke by increasing the flow of saliva, which can affect the species and relative abundance of oral opportunistic pathogens. In order to prove this, investigators need to (1) firstly conduct a randomized controlled trial to confirm whether hyperbaric oxygen therapy is able to reduce the levels of plaque, and the incidence of pneumonia complicating stroke at clinical level; (2) secondly employ metagenomics analysis to compare oral rinse samples and respiratory samples, and to identify pneumonia-associated "oral opportunistic pathogens group"; (3) finally elucidate how hyperbaric oxygen therapy influences the species and relative abundance of oral opportunistic pathogens. This proposed study will provide evidence for the integration of hyperbaric oxygen therapy as part of interdisciplinary stroke rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* New stroke events within 1-3 months (confirmed by CT and MRI)
* Moderate to severe disability (Barthel Index < 70)
* The patient is conscious, breathing autonomously, not undergoing tracheotomy or tracheal intubation for ventilator-assisted respiration
* No concurrent lower respiratory infections and other lung diseases
* The condition is relatively stable
* Cognitive function is normal to moderately impaired (Mini-Physical State Exchange, MMSE score>18)
* The Gugging Swallowing Screen (GUSS) shows swallowing difficulties
* No systemic and local use of antibiotic-containing mouthwash

Exclusion Criteria:

* A mild disability (Barthel Index > 70)
* The swallowing function is normal
* Indwelling nasogastric feeding tube
* The neurological status of the patient was significantly dynamically altered (significantly improved or worsened) in the short term prior to inclusion in the trial
* The patient had been treated with hyperbaric oxygen for other indications
* Had a chest condition and cannot withstand the pressure changes caused by hyperbaric oxygen therapy
* Have an inner ear disease
* Claustrophobia
* Communication barriers and inability to give informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of pneumonia | 2 months
  To calculate and compare the incidence of pneumonia between interventional group and control group, to identify whether the intervention approach could reduce the incidence.
Metagenomics | 2 months
  To analyze and compare the effect of intervention on the diversity of bacteria in saliva samples and lower respiratory sputum samples.

SECONDARY OUTCOMES:
Short Form Health Survey 12 (SF-12) | 2 months
  The concise health status scale (SF-12) IS used to assess the systemic health-related quality of life in stroke patients. It covers eight different areas: general health (GH), physical functioning (PF), bodily pain (BP), role-physical (RP), mental health (MH), vitality (VT), social functioning (SF), role-emotional (RE). The SF-12 consists of 12 items, and each of them has its own physical component summary (PCS) and mental component summary (MCS) regression coefficients. The response to each item will be multiplied by its PCS regression coefficient and added together with the PCS constant to provide Physical Health summary scores (SF-12 PCS). Mental Health summary scores (SF-12 MCS) will be calculated likewise. The higher the score, the higher the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Yinliang Qi, M.B.B.S., Study Director — The Second People's Hospital of Hefei
Locations (1):
- The Second People's Hospital of Hefei, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No